CLINICAL TRIAL: NCT02469610
Title: Assessment of Intercostal Block Scheduling in Preventing Acute Surgical and Post-surgical Pain in Thoracoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Dan Levy Faber, Dr, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMC-14-0123-CTIL
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Chest Pain; Surgery
Keywords: Post surgical pain
MeSH Terms: conditions — Chest Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- study (Experimental): In the study group the surgeon will perform an intercostal Bupivacaine block of 100ml over five intercostal spaces which include the operation cuts. The block will be done in the beginning of the surgery right after the insertion of the video camera to the pleural space.
  Interventions: Other: Intercostal block Bupivacaine based
- control (Other): In the control group the surgeon will perform the same intercostal block at the end of the surgery just before closing the operation cuts. this approach is used today in our department.
  Interventions: Other: Intercostal block Bupivacaine based

INTERVENTIONS:
Other: Intercostal block Bupivacaine based — Intercostal Bupivacaine block of 100ml over five intercostal spaces.

SUMMARY:
It is well known that chest surgery patients suffer from high level pain in the perioperative period. The transition to thoracoscopic approaches reduced surgical pain. The proper pain control technique for thoracoscopic approaches is still under debate. One of the most popular methods for pain control is these procedures is the Intercostal block. The Intercostal block is usually based upon topical analgesic. In this study the investigators will try to examine the effect on pain control of the timing of Intercostal block of 100 mg BUPIVACAINE. The study is a prospective comparative study. The cohort will be divided into two groups. In the control group patients will have Intercostal block after surgery and in the study group the intercostal block will be given in the beginning of the surgical procedure. All other analgesic treatment during and post-surgery will be the same in both groups. The study will evaluate pain level in the days after the surgery, analgesic medication consumption and relevant morbidity.

DETAILED DESCRIPTION:
Intercostal Bupivacaine block Intercostal block is a procedure during which a local anesthetic is injected to the intercostal space. This space includes the rote of the intercostal nerve. The purpose of the procedure is to block the neuropathic pain that developed due to inflammation and irritation of the nerve and other close structures. Some add steroids to the injection because of their anti-inflammatory effect.

Bupivacaine is a local anesthetic. It belongs to a group of medicines called amide- type local anesthetics. It is a well-known medication with many years of documented use in local and regional anesthesia. Bupivacaine binds to the intracellular portion of voltage-gated sodium channels and blocks sodium influx into nerve cells. This block prevents depolarization. The lack of depolarization precludes initiation or conduction of a pain signal can occur.

Study Aims This study will try to evaluate the difference in pain control during and post thoracoscopic surgery in patients who had bupivacaine intercostal block before versus after surgery.

The study main end point is the amount of analgesic medication consumption by patients during and after thoracoscopic surgery.

Secondary end points will include subjective patient's pain evaluation, length of hospital stay and post-operative complication.

Inclusion Criteria Thoracoscopic surgery candidate. Over 18 years old. No known allergy to Bupivacaine. Patient is able to read understand and singe an inform consent.

Exclusion Criteria Previous thoracic operation in the same side.

Study plan The study cohort will be divided into two groups. Study group and control group. Each group will include 30 thoracoscopic surgery candidates. The participants will be randomly assigned to the research groups using a computer selection done by the study team. The participants will not know as to which group they are assigned. All participants will by recruited in the cardio-thoracic surgery department, CARMEL medical center, Haifa, ISRAEL.

The basic thoracoscopic surgery approach uses three operation cuts the main Lateral surgical cut is less than 5 cm. Another lower cut of 1-2cmfor the video camera and a lateral subscapular cut of 1-2cm for lung retraction. No rib retractors are being used.

During surgery the anesthesiology team is in charge of patient sedation and analgesia according to the local anesthesia department protocol.

After surgery the thoracic team is in charge on patient analgesia treatment according to cardio-thoracic surgery department local protocol.

Patients will randomized into either study or control group. In the study group the surgeon will perform an intercostal Bupivacaine block of 100ml over five intercostal spaces which include the operation cuts. The block will be done in the beginning of the surgery right after the insertion of the video camera to the pleural space. In the control group the surgeon will perform the same intercostal block at the end of the surgery just before closing the operation cuts. All other operation stapes and analgesic treatment will be the same for both groups.

Follow up Patient follow up will include the perioperative hospitalization and will continue up to six months after discharge.

Follow up will include analgesic medication usage, pain levels, demographic details, Hospital length of stay, post-operative complication and time to resume daily routine.

ELIGIBILITY:
Inclusion Criteria:

* Thoracoscopic surgery candidate.
* Over 18 years old.
* No known allergy to Bupivacaine.
* Patient is able to read understand and singe an inform consent.

Exclusion Criteria:

* Previous thoracic operation in the same side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01-30 (Actual); Study Completion 2017-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CarmelMC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
general discricptive data only

REFERENCES:
- [Background] 1. Regional analgesia for video-assisted thoracic surgery: a systematic review.Steinthorsdottir KJ, Wildgaard L, Hansen HJ, Petersen RH, Wildgaard K. Eur J Cardiothorac Surg. 2013 Nov 27. 2. Postoperative analgesia in video-assisted thoracoscopy: the role of intercostal blockade. Taylor R, Massey S, Stuart-Smith K. J Cardiothorac Vasc Anesth. 2004 Jun;18(3):317-21. 3. The efficacy of intraoperative internal intercostal nerve block during video-assisted thoracic surgery on postoperative pain.Bolotin G, Lazarovici H, Uretzky G, Zlotnick AY, Tamir A, Saute M.Ann Thorac Surg. 2000 Dec;70(6):1872-5. 4. Preventing post-thoracotomy pain syndrome.Khelemsky Y, Noto CJ. Mt Sinai J Med. 2012 Jan-Feb;79(1):133-9. doi: 10.1002/msj.21286. Review. 5. Prevention of chronic pain after surgical nerve injury: amputation and thoracotomy.Buchheit T, Pyati S.Surg Clin North Am. 2012 Apr;92(2):393-407. Review. 6. Paravertebral blocks.Chelly JE. Anesthesiol Clin. 2012 Mar;30(1):75-90. Review. 7. Persistent postoperative pain: where are we now? Niraj G, Rowbotham DJ. Br J Anaesth. 2011 Jul;107(1):25-9. Review.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study | Control
Started | 34 | 31
Completed | 30 | 30
Not Completed | 4 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — exclusion criteria | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 7 | 20
  >=65 years | 17 | 23 | 40
Age, Continuous [Mean (Full Range); unit: years] | 64.6 [32 to 83] | 67.4 [23 to 86] | 66 [23 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 14 | 18 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Use
Description: The amount of analgesic medication consumption by patients during and after thoracoscopic surgery. the measurement include A. Analgesic usage during the hours of operation and recovery unit (4-8Hr) B. Analgesic usage during postoperative days (first, second, third and fourth for each 24 Hr)
Time Frame: post operative
Population: the use of opioids in the operative day (post operative day 0)
Measure: Mean (Standard Deviation); unit: MG
Arm/Group | Study | Control
Number analyzed (Participants) | 30 | 30
MG | 33.35 (10.31) | 35.32 (13.44)

2. Secondary Outcome: Visual Analog Pain Scale
Description: subjective patient's pain evaluation according to Visual Analog pain Scale (VAS). Visual Analog pain Scale a 1-10 score of pain. 1 being a lowest level of pain and 10 the worst pain felt by the patient.
Time Frame: post operative
Population: Visual Analog pain Scale on the first post-operative day. For each patient we calculate the average score of his answers to the question "How do you rate your pain on the Visual Analog pain Scale ?" during the first post-operative day.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study | Control
Number analyzed (Participants) | 30 | 30
units on a scale | 3.53 (2.64) | 3.63 (2.64)

ADVERSE EVENTS:
Time Frame: 1 months
Arm/Group | Study | Control
All-Cause Mortality (participants affected / at risk) | 1/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/31
Other Adverse Events (participants affected / at risk) | 0/34 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study (N=34) | Control (N=31)
massive pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT02469610/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT02469610/SAP_001.pdf
  • Informed Consent Form (2014-05-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT02469610/ICF_002.pdf